CLINICAL TRIAL: NCT03560154
Title: Effects of Whole Body Vibration Training in Patients With Interstitial Lung Disease: A Randomized Controlled Trial
Brief Title: Effects of Whole Body Vibration Training in Patients With Interstitial Lung Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Nur Selin Of, Principal Investigator, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N-85
Record Dates: First submitted 2018-06-06; First posted 2018-06-18 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Interstitial Lung Disease; Scleroderma; Idiopathic Pulmonary Fibrosis
Keywords: Pulmonary Function Test; Peripheral Muscle strength; Postural balance; Dyspnea; Pulmonary Muscle Strength; Functional Capacity; Fatigue; Quality of Life
MeSH Terms: conditions — Lung Diseases, Interstitial; Scleroderma, Diffuse; Idiopathic Pulmonary Fibrosis; Dyspnea; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Whole Body Vibration Training (Experimental): whole body vibration application will be performed in the range of 25-40 Hz, with amplitude 1-2 mm, 30-60 seconds (30-45 seconds) application and resting times of 60 seconds, 2-5 sets each session. In TVT training; Eight kinds of exercises will be provided, including 3 sessions per week for 4 weeks. The duration of each session will vary between 8-30 minutes. The frequency, amplitude, and duration of the TVT will be gradually increased from the lowest intensity to the level that the patient can tolerate. 8 exercises will be applied: for lower extremity; high squat, deep squat, right/left lunge, calf raise, for upper extremity; front raise, bent over lateral, biceps curl, and cross over. Before TVT application, 5-8 min. warm-up exercises will be applied. If desaturation (<88%) develops during the training in the patient, an oxygen mask will be used to ensure adequate oxygenation. Also, as a home program; respiratory exercises will be taught every day of the week for 10 minutes a day.
  Interventions: Other: Whole Body Vibration Training
- Home respiratory exercises (No Intervention): Respiratory exercises will be taught to the patient. Duration of the respiratory exercises is at least 10 minute per session, 7 days a week for 4 weeks. A weekly phone call will be provided and exercise will be followed.

INTERVENTIONS:
Other: Whole Body Vibration Training — whole body vibration application will be performed in the range of 25-40 Hz, with amplitude 1-2 mm, 30-60 seconds (30-45 seconds) application and resting times of 60 seconds, 2-5 sets each session. Also, as a home program; respiratory exercises will be taught every day of the week for 10 minutes a day.
  Arms: Whole Body Vibration Training

SUMMARY:
Interstitial lung disease (ILD) is a diverse group of parenchymal lung disorders characterized by restrictive lung function and impaired alveolar diffusion capacity, leading to dyspnea on exertion, reduced exercise endurance, and poor quality of life. Patients usually complain of progressive breathlessness, persisting non-productive cough, which occurs with exercise. Hemoptysis, fever, chest pain are also seen. The most common comorbidity in chronic lung diseases is the progressive loss of exercise tolerance. Not only dyspnea, but also peripheral muscle dysfunction and cognitive deficits such as, anxiety and depression are responsible for the reduction of mobility in the patient. In the context of pulmonary rehabilitation (PR) program to be applied in interstitial lung diseases; upper and lower limb endurance, stretching and relaxation techniques, aerobic exercise training, respiratory muscle training, training of energy conservation methods, support by determining oxygen requirement, nutritional evaluation, prevention of weight and muscle loss, psycho-social support. The purpose of PR programs in this disease is; to improve muscle strength, endurance, and mechanical activity, to improve dyspnea sensation, to improve functional capacity, to inform and educate the patient about the patient's disease. The use of whole body vibration (TVT) is an increasingly common method of therapeutic use in order to improve neuromuscular performance. TVT applications have shown that increases muscle activity, muscle strength and muscle strength, improves lower extremity blood circulation and balance, and increases growth hormone production. TVT training effects have rarely been studied in patients with pulmonary disease. Muscle strength and performance enhancement were significant effects of TVT, which was emphasized as a promising exercise method for those with chronic obstructive pulmonary disease (COPD). Over the past decade, endurance and strength training has been established as the most important components of exercise training programs in patients with COPD and ILD. Therefore, inclusion of TVT into exercise training programs in ILD patients may lead to beneficial results.

The investigators hypotheses are:

1. the combination of home respiratory exercises with whole body vibration training may lead to more improved respiratory muscle strength, dyspnoea, functional capacity, balance, peripheral muscle strength and quality of life in ILD patients
2. when applied as an isolated intervention, home respiratory exercises programme may lead to lower results than combination programs.

DETAILED DESCRIPTION:
Patients:

All participants with ILD will be recruited from a Cerrahpasa Medical Faculty Hospital between January 2017 and June 2018. All treatments will performed in the same hospital.

Sample Size:

"Power and Sample Size Program" was used to calculate sample size. Power analysis was done with Pass 11 Home program. In the power analysis program, α = 0,05, β = 0,15 1- β = 0,84. When the number of samples of the groups was 30 and 30, 84% power was obtained. Using a two-sided two-sample t-test, the standard deviations from the 0,05 alpha value are 7.0 and 6.0.

Procedure:

A list of individuals diagnosed with interstitial lung disease who are following the outpatient clinic of the Department of Chest Diseases of the Istanbul University Cerrahpaşa Medical Faculty and who meet the inclusion criteria for the study will be created. The created patient list will be enumerated. Two groups will be formed from the numbered persons by the random number table method (n = 60). Groups will receive 30 participants in the treatment group, whose protocol numbers end in an even number, and 30 members in the control group, who finished with an odd number of protocol numbers. Up to 10% of the sample size will be selected as a substitute, taking into account the non-participation of the selected individuals in the study.

Assessments at baseline and after training will be performed by pulmonary physiotherapist. All the participants will be treated in the Cerrahpaşa Medical Faculty hospital by a physiotherapist who is experienced in pulmonary rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with interstitial lung disease (Idiopathic Pulmonary Fibrosis, pneumoconiosis, chronic hypersensitivity pneumonia, radiation fibrosis, collagenosis pulmonary involvement, nonspecific interstitial pneumonitis-NSIP, idiopathic NSIP)
* Patients whose stability and medical treatment have not been changed for the last 3 months will be included in the study.

Exclusion Criteria:

* Malignant tumor,
* presence of co-morbidities that prevent exercise training (severe orthopedic or neurological deficit, unstable cardiac disease)
* The knee and / or hip joint replacement operation has been performed,
* having lower and upper limb amputation,
* taking any hormone replacement or medication that may affect the normal metabolism of the musculoskeletal system,
* presence of neurological (MS, intracranial tumor, neurodegenerative diseases, cerebrovascular event, epilepsy) disease which will affect balance and proprioception,
* those with drug use history (antidepressants, anticonvulsants, sedatives, betahistine) that may affect the balance,
* having Ischemic heart disease, dilate, hypertrophic or nonidiopathic cardiomyopathy,
* having pacemaker entity, By-pass, coronary stent,
* having uncontrolled DM,
* presence of acute arthritis / tendinopathy,
* O2 saturation in room air <80% (resting), patient with advanced respiratory failure,
* having severe neurological and / or metabolic pathologies,
* having hemodynamic instability,
* Being pregnant and breastfeeding,
* Individuals with a recent surgical operation, ILD, will not be included in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Pulmonary Function Test | 4 weeks
  The pulmonary function test (PFT) will be performed with a portable spirometry device (Spirobank II) with the nose closed and at least three times in the sitting position. After the nose is tightened with a latch, the person breathes normally on the spirometer. After a few normal inspirations and expirations, it is desirable to take a deep breath at the end of the expiration at the level of rest, and to release the air slowly and continuously afterwards. With this application, the volumes and capacities outside the residual volume (RV), functional residual capacity (FRC) and total lung capacity (TLC) are calculated.
Diffusing capacity for carbon monoxide (DLCO) | 4 weeks
  The single breath carbon monoxide diffusion test method will be used to calculate the diffusion capacity. Carbonmonoxide Diffusion (DLCO) measurement is an important noninvasive test that provides information on pulmonary gas exchange. The CO concentrations are measured by passing the analyzer through a breathing air analyzer of the patient, which is then exhaled into the device; the amount of CO transferred to the blood is calculated from the difference between the inspired air and the CO concentrations in the expired air.
Respiratory muscle strength | 4 weeks
  Respiratory muscle strength will be measured using a portable electronic mouth measuring instrument (MicroRPM; Micro Medical, UK). Maximum inspiratory (MIP) and expiratory (MEP) pressures are noninvasive tests that indirectly indicate respiratory muscle strength. It is the intraoral pressure measured during maximal inspiration and maximal respiration against a valve (shutter) that closes the respiratory tract during expiration. The best of three measurements is accepted.
6-minute walk test (6MWT) | 4 weeks
  Functional exercise capacity was assessed using the 6-minute walk test (6MWT). Patients will be walked in a 30-meter-long corridor for 6 minutes and the maximum walking distance will be measured. Before and after the test, heart rate, blood pressure and pulse oximeter will measure O2 saturation, and according to Borg scale, dyspnea and fatigue level will be determined. Oxygen will be provided immediately following exercise for patients who desaturate (SpO2 <88%), or as needed.
6-minute pegboard and ring test (6PBRT) | 4 weeks
  Subjects are asked to sit straight in a chair and a pegboard with multiple peg positions is placed in front of the subject at arm's length from the body. Two pegs are positioned at the shoulder level and 2 at 20 cm above the shoulder level, and 10 rings (1/2 oz per ring) are put on each of the 2 lower pegs. The final score is the total number of rings moved during the 6-minute period. Subjects are permitted to stop and rest during the test if they feel severe dyspnea, fatigue, or other discomfort, and continue moving the pegs as soon as they can. Subjects are asked to score the perceived dyspnea and fatigue after the test by the Borg scale. Each subject performe the PBRT twice. A pulse oximeter is used to monitor heart rate (HR) and arterial oxygen saturation (Sao2), and measure blood pressure (BP) before and after each test.

SECONDARY OUTCOMES:
Timed Up and Go Test (TUG) | 4 weeks
  TUG is a reliable and simple test to assess balance and functional mobility of stroke patients. The patient sited in chair and with command of physiotherapist raised from the chair, walked 3 meters, walked back to the chair and sited down again. The time of process was recorded by the physiotherapist in seconds. It was allowed to use walking aid during the test. Lower duration indicates better mobility performance.
Sit to Stand Test (STS) | 4 weeks
  It is a test based on crossing the patient's hands at the chest and making the most repetition possible by sitting and lifting continuously for 30 seconds. The number of sit down and stand up is recorded by the physiotherapist.
Static Posturography System (TETRAX) | 4 weeks
  Static posturography formed with four separate plates and each force plate measures the perpendicular pressure of the anterior and posterior feet. Subjects took off their shoes, positioned their feet on the plates, and stood in a comfortable position. Eight different postures were evaluated for the test and each posture was measured for 32 seconds. For the postural variable factors, the stability index (ST), Fourier index, weight distribution index (WDI), and the synchronization index (SI) are measured.
Peripheral Muscle Strength Measurement | 4 weeks
  Quadriceps femoris and biceps brachii isometric muscle strength will be measured by portable hand dynamometer (JTECH, Medical Commander Powertrack II, USA). Isometric muscle strength of Quadriceps femoris and biceps brachii is measured by portable hand dynamometer. Quadriceps femoris muscle force is measured in sitting position, at knee extension, and biceps brachii muscle strength at backrest position, while elbow is flexed. The measurements are repeated three times in succession and the average is recorded.
The Fatigue Severity Scale (FSS) | 4 weeks
  The Fatigue Severity Scale is a self-administered questionnaire with 9 items (questions) investigating the severity of fatigue in different situations during the past week. Respondents answer using a Likert scale ranging from 1 to 7. ''1'' indicates strong disagreement with the statement, while ''7'' indicates strong agreement. Total score is calculated by deriving an arithmetic mean. FSS scores range from 0-63. A score of 36 or higher generally indicates severe fatigue.
St. George's Respiratory Questionnaire (SGRQ) | 4 weeks
  The SGRQ is a standardized self-administered airways disease-specific questionnaire. It contains 50 items (covering 76 levels) divided into three subscales: ''Symptoms'' (8 items), including several respiratory symptoms, their frequency and severity; ''Activity'' (16 items), concerned with activities that cause or are limited by breathlessness; and ''Impacts'' (26 items), which covers a range of aspects concerned with social functioning and psychological disturbances resulting from airways disease. SGRQ scores range from 0-100, zero score indicating no impairment of life quality. Answers to SGRQ items are weighted and total SGRQ score and scores on the three subscales (Symptom frequency, Impact, and Activity) are calculated by adding these weights. Scores are then converted to percentages by dividing the weighted score obtained by the total possible weighted score. The higher the score the poorer the quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Zerrin Yiğit, Prof, Study Director — Istanbul University/Institute of Cardiology
Locations (1):
- Nur Selin Of, Istanbul, Istanbul University/Cerrahpasa Faculty of Medicine, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Salhi B, Malfait TJ, Van Maele G, Joos G, van Meerbeeck JP, Derom E. Effects of Whole Body Vibration in Patients With COPD. COPD. 2015;12(5):525-32. doi: 10.3109/15412555.2015.1008693. Epub 2015 Aug 4. PMID 26457458
- [Background] Turner S, Torode M, Climstein M, Naughton G, Greene D, Baker MK, Fiatarone Singh MA. A randomized controlled trial of whole body vibration exposure on markers of bone turnover in postmenopausal women. J Osteoporos. 2011;2011:710387. doi: 10.4061/2011/710387. Epub 2011 Jun 27. PMID 21772975
- [Background] Gloeckl R, Jarosch I, Bengsch U, Claus M, Schneeberger T, Andrianopoulos V, Christle JW, Hitzl W, Kenn K. What's the secret behind the benefits of whole-body vibration training in patients with COPD? A randomized, controlled trial. Respir Med. 2017 May;126:17-24. doi: 10.1016/j.rmed.2017.03.014. Epub 2017 Mar 14. PMID 28427544
- [Background] Gloeckl R, Heinzelmann I, Kenn K. Whole body vibration training in patients with COPD: A systematic review. Chron Respir Dis. 2015 Aug;12(3):212-21. doi: 10.1177/1479972315583049. Epub 2015 Apr 22. PMID 25904085
- [Background] Cardim AB, Marinho PE, Nascimento JF Jr, Fuzari HK, Dornelas de Andrade A. Does Whole-Body Vibration Improve the Functional Exercise Capacity of Subjects With COPD? A Meta-Analysis. Respir Care. 2016 Nov;61(11):1552-1559. doi: 10.4187/respcare.04763. Epub 2016 Sep 20. PMID 27651524
- [Background] Polatli M, Yorgancioglu A, Aydemir O, Yilmaz Demirci N, Kirkil G, Atis Nayci S, Kokturk N, Uysal A, Akdemir SE, Ozgur ES, Gunakan G. [Validity and reliability of Turkish version of St. George's respiratory questionnaire]. Tuberk Toraks. 2013;61(2):81-7. doi: 10.5578/tt.5404. Turkish. PMID 23875584
- [Background] Deniz S, Sahin H, Yalniz E. Does the severity of interstitial lung disease affect the gains from pulmonary rehabilitation? Clin Respir J. 2018 Jun;12(6):2141-2150. doi: 10.1111/crj.12785. Epub 2018 Mar 24. PMID 29498799
- [Background] Dowman L, Hill CJ, Holland AE. Pulmonary rehabilitation for interstitial lung disease. Cochrane Database Syst Rev. 2014 Oct 6;(10):CD006322. doi: 10.1002/14651858.CD006322.pub3. PMID 25284270
- [Background] Hanada M, Sakamoto N, Ishimatsu Y, Kakugawa T, Obase Y, Kozu R, Senjyu H, Izumikawa K, Mukae H, Kohno S. Effect of long-term treatment with corticosteroids on skeletal muscle strength, functional exercise capacity and health status in patients with interstitial lung disease. Respirology. 2016 Aug;21(6):1088-93. doi: 10.1111/resp.12807. Epub 2016 May 13. PMID 27173103
- [Background] Schaeffer MR, Ryerson CJ, Ramsook AH, Molgat-Seon Y, Wilkie SS, Dhillon SS, Mitchell RA, Sheel AW, Khalil N, Camp PG, Guenette JA. Neurophysiological mechanisms of exertional dyspnoea in fibrotic interstitial lung disease. Eur Respir J. 2018 Jan 18;51(1):1701726. doi: 10.1183/13993003.01726-2017. Print 2018 Jan. PMID 29348183
- [Background] Nishiyama O, Yamazaki R, Sano H, Iwanaga T, Higashimoto Y, Kume H, Tohda Y. Physical activity in daily life in patients with idiopathic pulmonary fibrosis. Respir Investig. 2018 Jan;56(1):57-63. doi: 10.1016/j.resinv.2017.09.004. Epub 2017 Oct 23. PMID 29325683
- [Background] Yilmaz Yelvar GD, Cirak Y, Dalkilinc M, Demir YP, Baltaci G, Komurcu M. Impairments of postural stability, core endurance, fall index and functional mobility skills in patients with patello femoral pain syndrome. J Back Musculoskelet Rehabil. 2017;30(1):163-170. doi: 10.3233/BMR-160729. PMID 27392843
- [Background] Akkaya N, Doganlar N, Celik E, Aysse SE, Akkaya S, Gungor HR, Sahin F. TEST-RETEST RELIABILITY OF TETRAX(R) STATIC POSTUROGRAPHY SYSTEM IN YOUNG ADULTS WITH LOW PHYSICAL ACTIVITY LEVEL. Int J Sports Phys Ther. 2015 Nov;10(6):893-900. PMID 26618068
- [Background] Wickerson L, Mathur S, Helm D, Singer L, Brooks D. Physical activity profile of lung transplant candidates with interstitial lung disease. J Cardiopulm Rehabil Prev. 2013 Mar-Apr;33(2):106-12. doi: 10.1097/HCR.0b013e3182839293. PMID 23403914
- [Background] Dale MT, McKeough ZJ, Munoz PA, Corte P, Bye PT, Alison JA. Physical activity in people with asbestos related pleural disease and dust-related interstitial lung disease: An observational study. Chron Respir Dis. 2015 Nov;12(4):291-8. doi: 10.1177/1479972315587518. Epub 2015 Jun 5. PMID 26048393
- [Background] Dale MT, McKeough ZJ, Troosters T, Bye P, Alison JA. Exercise training to improve exercise capacity and quality of life in people with non-malignant dust-related respiratory diseases. Cochrane Database Syst Rev. 2015 Nov 5;2015(11):CD009385. doi: 10.1002/14651858.CD009385.pub2. PMID 26544672
- [Background] Dowman L, McDonald CF, Hill C, Lee A, Barker K, Boote C, Glaspole I, Goh N, Southcott A, Burge A, Ndongo R, Martin A, Holland AE. The benefits of exercise training in interstitial lung disease: protocol for a multicentre randomised controlled trial. BMC Pulm Med. 2013 Feb 1;13:8. doi: 10.1186/1471-2466-13-8. PMID 23369075
- [Background] Tonelli R, Cocconcelli E, Lanini B, Romagnoli I, Florini F, Castaniere I, Andrisani D, Cerri S, Luppi F, Fantini R, Marchioni A, Beghe B, Gigliotti F, Clini EM. Effectiveness of pulmonary rehabilitation in patients with interstitial lung disease of different etiology: a multicenter prospective study. BMC Pulm Med. 2017 Oct 10;17(1):130. doi: 10.1186/s12890-017-0476-5. PMID 29017478
- [Background] Janaudis-Ferreira T. Exercise training improves exercise capacity and quality of life in people with interstitial lung disease [synopsis]. J Physiother. 2017 Oct;63(4):257. doi: 10.1016/j.jphys.2017.07.002. Epub 2017 Sep 6. No abstract available. PMID 28888691
- [Background] Wickerson L. Exercise training improves exercise capacity and quality of life in people with interstitial lung disease [commentary]. J Physiother. 2017 Oct;63(4):257. doi: 10.1016/j.jphys.2017.07.001. Epub 2017 Sep 6. No abstract available. PMID 28888689
- [Background] Keyser RE, Christensen EJ, Chin LM, Woolstenhulme JG, Drinkard B, Quinn A, Connors G, Weir NA, Nathan SD, Chan LE. Changes in fatigability following intense aerobic exercise training in patients with interstitial lung disease. Respir Med. 2015 Apr;109(4):517-25. doi: 10.1016/j.rmed.2015.01.021. Epub 2015 Feb 7. PMID 25698651
- [Background] Caron M, Hoa S, Hudson M, Schwartzman K, Steele R. Pulmonary function tests as outcomes for systemic sclerosis interstitial lung disease. Eur Respir Rev. 2018 May 15;27(148):170102. doi: 10.1183/16000617.0102-2017. Print 2018 Jun 30. PMID 29769294
- [Background] Szentes BL, Kreuter M, Bahmer T, Birring SS, Claussen M, Waelscher J, Leidl R, Schwarzkopf L. Quality of life assessment in interstitial lung diseases:a comparison of the disease-specific K-BILD with the generic EQ-5D-5L. Respir Res. 2018 May 25;19(1):101. doi: 10.1186/s12931-018-0808-x. PMID 29801506
- [Background] Ramadurai D, Riordan M, Graney B, Churney T, Olson AL, Swigris JJ. The impact of carrying supplemental oxygen on exercise capacity and dyspnea in patients with interstitial lung disease. Respir Med. 2018 May;138:32-37. doi: 10.1016/j.rmed.2018.03.025. Epub 2018 Mar 26. PMID 29724390
- [Background] Suzuki A, Kondoh Y, Swigris JJ, Ando M, Kimura T, Kataoka K, Yamano Y, Furukawa T, Numata M, Sakamoto K, Hasegawa Y. Performance of the St George's Respiratory Questionnaire in patients with connective tissue disease-associated interstitial lung disease. Respirology. 2018 Mar 25. doi: 10.1111/resp.13293. Online ahead of print. PMID 29575410